CLINICAL TRIAL: NCT02666300
Title: To Compare the Incidence of Postoperative Sore Throat Between a TaperGuardEndotracheal Tube(ETT)and a Cylindrical-shaped ETT Under Highcuffpressure:A Randomized,Double-blindTrial.
Brief Title: To Compare the Incidence of POST Between a TaperGuard ETT and Cylindrical-shaped ETT Under High Cuff Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: post2015taper
Record Dates: First submitted 2016-01-18; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Postoperative Complications
Keywords: Postoperative sore throat,Anesthesia
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TaperGuard ETT (Experimental): tracheal intubation with the TaperGuard ETT，the ETT cuff is Taper-shangped.
  Interventions: Other: TaperGuard ETT

INTERVENTIONS:
Other: TaperGuard ETT — tracheal intubation with TaperGuard ETT

SUMMARY:
Postoperative Sore Throat (POST) is supposed to be the most frequently occurred respiratory complication related to endotracheal intubation .Whether the new type of ETT(TaperGuard ETT) to decrease or to increase the complications of general anesthesia compared with Cylindrical-shaped ETT is still unknown .In this study ,we will compare the different incidence of complications following general anesthesia between TaperGuard ETT and Cylindrical-shaped ETT under high endotracheal tube cuff pressure.

DETAILED DESCRIPTION:
BACKGROUND:Postoperative Sore Throat (POST) is supposed to be the most frequently occurred respiratory complication related to endotracheal intubation .Endotracheal tube size ,airway manipulation ,patients position et al. have been recognized as the factors affecting Postoperative Sore Throat .Controversy in respect of the relationship between the cuff design and POST is still existed. Whether the new type of ETT (TaperGuard ETT) to decrease or to increase the complications of general anesthesia compared with Cylindrical-shaped ETT is still unknown .In this study ,we will compare the different incidence of complications following general anesthesia between TaperGuard ETT and Cylindrical-shaped ETT under high endotracheal tube cuff pressure.

METHODS:Patients undergoing elective non-throat and non-neck surgery were randomly allocated to receive either a TaperGuard ETT(group T) or Cylindrical-shaped ETT ( Group C).Patients received general anesthesia with different endotracheal tubes .Recoil of inflation syringe plunger was used to inflate the cuff. In the study , the cuff pressures of the endotracheal tube were recorded by a calibrated cuff manometer at two time: when the intubation was complited and before endotracheal tube was removed. The incidence and severity of Postoperative Sore Throat(POST),hoarseness, cough were collected by a single investigator blinded to the experiment at 0, 1,6, 12, and 24 hours post-operation.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia surgery

aged 18 to 75 years

ASA classⅠ or Ⅱ

undergoing elective non-throat and non-neck surgery under generalanesthesia

intubation timemore than two hours

BMI≤30 kg／m2

Exclusion Criteria:

* Patients with ahistory of preoperative sore throat

known airway disease and difficult intubation

more than one attempt at intubation

Mallampati grade 3 to 4

Cormack-Lehane grade3 to 4

BMI >35 Kg/m2

Those have an operation with the lateral flank or prone position

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of Participants with TaperGuard ETT at 0,1,,6,12,24 hours post-operative | 0,1,,6,12,24 hours post-operative
The incidence and severity of Participants with Cylindrical ETT at 0,1,,6,12,24 hours post-operative | 0,1,,6,12,24 hours post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Z Yang, MD,PhD, Principal Investigator — The Second Affiliated Hospital of Dalian Medical University
Locations (1):
- The Second Hospital of Dalian Medical University, Dalian, Liaoning, China